CLINICAL TRIAL: NCT01234779
Title: A Phase II, Multi-center, Randomized, 4-week, Double-blind, Parallel Group, Placebo and Active-controlled Trial of the Safety and Efficacy of RO4917838 vs. Placebo in Patients With an Acute Exacerbation of Schizophrenia
Brief Title: A Study of RO4917838 (Bitopertin) in Patients With Acute Exacerbation of Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WN25333; 2010-021984-33
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — (4-(3-fluoro-5-trifluoromethylpyridin-2-yl)piperazin-1-yl)(5-methanesulfonyl-2-(2,2,2-trifluoro-1-methylethoxy)phenyl)methanone; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- A (Experimental)
  Interventions: Drug: bitopertin [RO4917838]
- B (Experimental)
  Interventions: Drug: bitopertin [RO4917838]
- C (Active Comparator)
  Interventions: Drug: olanzapine
- D (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bitopertin [RO4917838] — 10 mg orally daily, 4 weeks
  Arms: A
Drug: bitopertin [RO4917838] — 30 mg orally daily, 4 weeks
  Arms: B
Drug: olanzapine — 15 mg orally daily, 4 weeks
  Arms: C
Drug: placebo — orally daily, 4 weeks
  Arms: D

SUMMARY:
This randomized, double-blind, placebo- and active-controlled, parallel group study will evaluate the safety and efficacy of RO4917838 (bitopertin) in patients with acute exacerbation of schizophrenia. Patients will be randomized to receive either RO4917838 10 mg or RO4917838 30 mg or olanzapine 15 mg or placebo orally daily for 4 weeks as inpatients, with a 4-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18-65 years of age
* Diagnosis of schizophrenia (Diagnostic and Statistical Manual of Mental Disorders DSM IV-TR)
* Acute exacerbation which began within the prior 8 weeks
* Female patients must be surgically sterile or post-menopausal, or agree to use effective contraception for the duration of the study

Exclusion Criteria:

* Current psychiatric diagnosis other than schizophrenia
* Alcohol or substance dependence within 3 months or abuse within 1 month (except for nicotine)
* Electro-convulsive therapy (ECT) within the prior 6 months
* Previous treatment with RO4917838 or another GLYT inhibitor
* Current treatment with olanzapine, or previous treatment with intolerability or lack of response
* Treatment with long-acting injectable antipsychotic within 2 dosing intervals
* Treatment with > 2 antipsychotics within 3 months
* History of neuroleptic malignant syndrome
* Have treatment-resistant schizophrenia as judged by treating physician or have failed two trials according to criteria in protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2011-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Syndrome Scale (PANSS) total score | from baseline to Day 28
Safety: Incidence adverse events | 8 weeks

SECONDARY OUTCOMES:
Clinical response, defined as at least 30% or 50% improvement from baseline PANSS total score | from baseline to Day 28
Change in symptomatology as measured by the PANSS factor and subscale scores | from baseline to Day 28
Global improvement as measured by the Clinical Global Impressions-Severity (CGI-S) scale | from baseline to Day 28
Global improvement as measured by the Clinical Global Impressions-Change (CGI-C) rating scale | from baseline to Day 28
Observable behavioural change as determined by the Nurses' Observation Scale For Inpatient Evaluation (NOSIE) | from baseline to Day 28
Time to readiness for discharge from inpatient unit as assessed by the Readiness For Hospital Discharge Questionnaire (RDQ) | from baseline to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (39):
- United States (19):
  - Little Rock, Arkansas
  - Cerritos, California
  - Oceanside, California
  - Pico Rivera, California
  - San Diego, California
  - Lauderhill, Florida
  - North Miami, Florida
  - Atlanta, Georgia
  - Lake Charles, Louisiana
  - Flowood, Mississippi
  - St Louis, Missouri
  - Willingboro, New Jersey
  - Holliswood, New York
  - New York, New York
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Charlesston, South Carolina
  - Austin, Texas
  - Irving, Texas
- Romania (5):
  - Arad
  - Bucharest
  - Foscani
  - Oradea
  - Târgovişte
- Russia (5):
  - Gatchina
  - Moscow
  - Petrozavodsk
  - Saint Petersburg
  - Talagi
- Slovakia (4):
  - Bojnice
  - Bratislava
  - Liptovský Mikuláš
  - Michalovce
- Ukraine (6):
  - Dnipropetrovsk
  - Donetsk
  - Kherson,Vil. Stepanivka
  - Kyiv
  - Poltava
  - Vinnytsia